CLINICAL TRIAL: NCT02382510
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Two-Way Cross-Over, Phase 2a Study to Evaluate the Safety and Bronchodilator Activity of TRN-157 in Stable Mild and Moderate Asthmatics
Brief Title: Multiple Ascending Dose Study of TRN-157 in Stable Mild and Moderate Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theron Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TRN-157-102
Record Dates: First submitted 2015-02-17; First posted 2015-03-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- TRN-157 (Experimental)
  Interventions: Drug: TRN-157
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: TRN-157
  Arms: TRN-157
Other: Placebo
  Arms: Placebo
Drug: Tiotropium
  Arms: Tiotropium

SUMMARY:
This multiple ascending dose study is to determine the safety and bronchodilator activity of TRN-157 in 59 mild and moderate asthmatics.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria will be considered eligible to participate in the study:

* The patient is ≥ 18 and < 70 years of age, and gives informed consent
* Clinical diagnosis of mild to moderate asthma of at least 6 months duration and age of onset < 50 years
* Presently using ICS at moderate doses (equivalent to 200-800 µg of budesonide or 88-500 µg of fluticasone daily)
* ≥ 12% and ≥ 200 mL improvement in FEV1 to 4 puffs albuterol by metered-dose inhaler (MDI) at screening visit
* Patient is willing to use acceptable form of birth control during trial and for one month thereafter
* Ability to measure morning (AM) peak expiratory flow (PEF) on schedule using electronic peak flow meter (EPFM) and to complete the study diary correctly at least 70% of the time during the run-in period
* After 7 day withdrawal from LABA therapy and overnight withdrawal from SABA therapy (except rescue medication), patient has between 55% - 80% of predicted FEV1 at CV2

Exclusion Criteria:

A patient meeting any of the following criteria is not eligible for enrollment in the study:

* A clinical diagnosis of chronic obstructive pulmonary disease (COPD), chronic bronchitis, bronchiectasis, or other significant pulmonary disease other than asthma
* History of upper or lower respiratory infection within 4 weeks of screening
* History of asthma exacerbation requiring oral or systemic corticosteroids or hospital admission within 6 months of screening
* History of myocardial infarction, or cardiac conduction abnormalities, including but not limited to atrial fibrillation, and paroxysmal atrial tachycardia
* Hospitalization due to cardiac failure within the last 6 months
* History of narrow angle glaucoma or obstructive uropathy
* Current smokers or vapers, or former smokers with > 10 pack-year (self-reported) history of smoking
* Patients who presently use the following medications will not be eligible for participation:

  * Long-acting muscarinic receptor antagonist (LAMA)
  * LABA (but may be withdrawn and converted to SABA x 7 days prior to entry)
  * Leukotriene pathway blockers
  * Anti-IgE antibody (Xolair) within last 6 months prior to CV1
  * Phosphodiesterase 4 (PDE4) inhibitors (e.g., Roflumilast)
  * Cromolyn
  * Methylxanthines (e.g., aminophylline and theophylline)
  * 5-Lipoxygenase inhibitor (e.g., Zileuton)
* Allergies to LAMA therapies
* History of life-threatening asthma exacerbation requiring ICU admission, mechanical ventilation, or tracheostomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FEV1 | After 2 weeks of treatment with TRN-157 vs. Placebo
Safety and tolerability as determined by number of subjects with adverse events | After 2 weeks of treatment with TRN-157 vs. Placebo
  Adverse events and/or clinically significant changes in vital signs, ECG, and/or laboratory values

SECONDARY OUTCOMES:
Characterize effects on pulmonary function | After 2 weeks of treatment with TRN-157 vs. Placebo
  FEV1(0-4 h); FVC AUC(0-4 h); FVC(0-4 h); Morning PEFR; Trough (pre-dose) FEV1
Characterize effects on asthma symptomatology | During the 2 weeks of treatment with TRN-157 vs. Placebo
  Asthma symptoms, including exacerbations; Number of asthma-control days; Rescue inhaler use; Nocturnal symptoms
Determination of pharmacokinetic parameters: AUC0-t, AUC0-inf, Cmax, tmax, t½, elimination rate constant (kel), volume of distribution at steady state (Vss/F), total plasma clearance (CL/F) | After 2 weeks of treatment with TRN-157
  AUC0-t, AUC0-inf, Cmax, tmax, t½, elimination rate constant (kel), volume of distribution at steady state (Vss/F), total plasma clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Krantz, MD, PhD, Study Director — Theron Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - WCCT Global, Costa Mesa, California
  - Allied Clinical Research, Gold River, California
  - Allied Clinical Research, Reno, Nevada
  - Dr. Winder & Associates/Toledo Center for Clinical Research, Sylvania, Ohio
  - The Allergy and Asthma Center of Southern Oregon, Medford, Oregon
  - West Houston Clinical Research Services, Houston, Texas
  - Sylvana Research, San Antonio, Texas